CLINICAL TRIAL: NCT04741464
Title: Effect of Tinzaparin on Inflammatory Biomarkers During the Acute Phase of Deep Vein Thrombosis
Acronym: Aticks Live
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0142
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Deep Vein Thrombosis; Inflammatory Response
Keywords: Deep Vein Thrombosis; Inflammatory Response
MeSH Terms: conditions — Venous Thrombosis | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tinzaparin — Tinzaparin 20 000 anti-Xa IU/mL dispensed in graduated syringes of 0.5 mL, 0.7 mL and 0.9 mL at the dose of 175IU/Kg/d.
  Strategy: Tinzaparin 175 UI/Kg/d for 21 days After this time the physician will continue the treatment of his choice to treat DVT.

SUMMARY:
Anticoagulants influence either coagulation, inflammation and inflammatory processes in deep vein thrombosis (DVT). Acute DVT cause an inflammatory response that may persist for a long period of time. There is a need to describe patterns of change in serum biomarker levels after acute DVT, and explore the association between trajectory biological patterns and clinical evolution in the era of various anticoagulants in the acute phase of treatment in order to be able to further avoid recurrence and late sequelae. It appears that direct oral anticoagulants and heparin alter inflammatory markers in different ways. It is therefore important to study the evolution of markers according to the different treatments used and secondarily to compare them with each other. Tinzaparin is used in the long term in patients with DVT, it is necessary to measure the evolution of inflammatory markers and then in another study to compare with the other molecules.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a first episode of symptomatic, proximal DVT of the lower limbs, confirmed by Duplex Ultrasound (DUS)
* Indication for treatment with Tinzaparin
* Patient covered by French national health insurance,
* Written informed consent.

Exclusion Criteria:

* Recent DVT (less than 2 months) objectively proven by venous ultrasound - Severe ilio-femoral DVT requiring recanalization
* Duration of treatment of more than 24 h since diagnosis
* Patients with acute symptoms (leg pain and swelling) for more than 5 days
* Planned surgery in the following 3 weeks, impossible to postpone
* Active haemorrhage or high risk of haemorrhage
* Symptoms of Post Thrombotic Syndrome
* Active neoplasm
* APL syndrome
* Renal insufficiency (Creatinine clearance (Cockcroft-Gault) <20 mL/min)
* Hepatic disease / or Hepatic Insufficiency / or serious liver disease
* Hyperkaliemia more than 5 mmol/L
* Patients with mechanical prosthetic heart valve
* weight more than 105 kgs in order to avoid difficulties with a dosage of 20000UI OF TINZAPARIN Any anti-inflammatory drugs or anti-platelet therapy
* Any other concomitant anticoagulant treatment such as VKA, heparin, fondaparinux and direct oral anticoagulants
* Contraindications to tinzaparin according to their SmPC
* Patient with asthma, If patients need to receive tinzaparin 10000UI antiX-a/0.5ml for the study,(due to sodium metabisulfite in the solution)
* Pregnant women or breastfeeding
* patient with age under 18
* Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
I-CAM levels variation in acute DVT patient | one year
  The main objective of the present study is to illustrate the I-CAM serum levels decrease after an acute DVT.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No